CLINICAL TRIAL: NCT03540342
Title: Evaluation of the Strategy of "One-stop" Endovascular Treatment for Concomitant Coronary Artery Disease and Aortic Atherosclerotic Disease
Brief Title: Evaluation of One-stop Strategy of EVAR and PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yi-Da Tang, Clinical professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z171100000417021
Record Dates: First submitted 2018-04-11; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Aortic Atherosclerotic Disease
Keywords: coronary artery disease; aortic atherosclerotic disease; one-stop; percutaneous coronary intervention; endovascular aortic repair
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One stop strategy group (Experimental): Percutaneous coronary intervention (PCI) will be performed on the same operating table immediately after the endovascular aortic repair (EVAR)
  Interventions: Procedure: One stop strategy group
- Staging strategy group (No Intervention): PCI will be performed several days after EVAR

INTERVENTIONS:
Procedure: One stop strategy group — Percutaneous coronary intervention (PCI) will be performed on the same operating table immediately after the endovascular aortic repair (EVAR)
  Arms: One stop strategy group

SUMMARY:
The study is designed to evaluate the safety and effectiveness of the "one-stop" endovascular intervention strategy for patients with concomitant coronary artery disease and aortic atherosclerotic disease. It is a registration study, which will consecutively enroll at least 50 patients with at least 30 subjects receiving one-stop strategy.

DETAILED DESCRIPTION:
It is a registration study, at least 50 patients will be consecutively enrolled and then be allocated into one-stop strategy group or staging strategy group with at least 30 subjects receiving one-stop strategy. In one stop strategy group, percutaneous coronary intervention (PCI) will be performed on the same operating table immediately after the endovascular aortic repair (EVAR). In staging strategy group, PCI will be performed several days after EVAR. The safety and effectiveness will be assessed between the two groups untill 1 year after the operation. The economic index will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years to 75years, male or female;
* Aortic atherosclerotic disease with the indication of EVAR;
* Coronary heart disease with the indication of PCI;
* Provided informed consent.

Exclusion Criteria:

* Acute aortic dissection
* Acute coronary syndrome
* Dysfunction of coagulation system
* Patients with gastrointestinal hemorrhage
* Known allergy to contrasts or antiplatelet drugs
* Renal dysfunction (GFR≤60ml/min)
* Patient with multi-branch coronary preferred CABG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events | 12 months
  The incidence of a composite endpoint of all-cause mortality, myocardial infarction, rupture of aorta, hematoma, bleeding events (BARC≥2 grade), pseudoaneurysm, stent thrombosis

SECONDARY OUTCOMES:
Operative success rate | 12 months
Average in-patient time | 12 months
Average cost during hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China